CLINICAL TRIAL: NCT03906708
Title: Physiological Phenotyping of Respiratory Outcomes in Infants Born Premature
Acronym: P3
Status: Active, not recruiting | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Robert Tepper, Professor of Pediatrics, MD, PhD, Indiana University
Other Study IDs: 1809404763; 1R01HL145679-01A1 (NIH)
Record Dates: First submitted 2019-03-18; First posted 2019-04-08 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Premature Lungs
MeSH Terms: interventions — Carbon Monoxide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Proteomics analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Premature Infants: Premature infants born between 24+0 and 36+6 weeks of gestation.
  Interventions: Other: Diffusion Capacity of the Lung for Carbon Monoxide (DLCO)

INTERVENTIONS:
Other: Diffusion Capacity of the Lung for Carbon Monoxide (DLCO) — Infant lung function testing

SUMMARY:
The purpose of this study is to examine if infants are more likely to suffer from respiratory complications during their first year of life due to being born premature.

DETAILED DESCRIPTION:
The overall objective of this study is to determine if infant respiratory morbidities after preterm birth are highly variable due to differential impairment of airway, parenchymal and vascular development that can be characterized as distinct physiologic phenotypes. If the nature and severity of these specific impairments of lung function are strongly associated with increased respiratory morbidities during infancy and that proteomic biomarkers can enhance the physiologic characterization of phenotype and prediction of late respiratory outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Infants born to mothers who are between the gestational ages of 24+0 and 36+6 weeks.

Exclusion Criteria:

* Cardiopulmonary defects
* Chromosomal defects
* Structural abnormalities of the upper airway, chest wall, or lungs
* Neurological/Neuromuscular disorders
* Infant not considered viable
* Family unlikely to be available for long term follow up
* Mothers under the age of 18.
* Non English speaking

Ages: 24 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Recruiting infants born between 24+0 and 36+6 weeks gestational age
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Infant lung development measured by diffusion lung capacity (DLCO). | By 5 months CGA.
  To characterize respiratory phenotypes through specific physiologic measures that quantify and identify predominant small airways, parenchymal and vascular dysfunction at 4 months CA and determine whether these phenotypes define risks for late respiratory morbidity during infancy.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Tepper, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Jeff Bjerregaard, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided